CLINICAL TRIAL: NCT03399942
Title: Treatment of Chronic Refractory Pain by Combined Deep Brain Stimulation of the Anterior Cingulum and Sensory Thalamus: a Feasibility and Safety Study
Brief Title: Combined Cingulate and Thalamic DBS for Chronic Refractory Chronic Pain
Acronym: EMOPAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 16-AOIP-01
Record Dates: First submitted 2017-12-01; First posted 2018-01-17 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Chronic Refractory Neuropathic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBS-ACC ON (Experimental): Start of stimulation of the DBS-ACC: On the first period, between M4 and M7, the DBS-ACC is ON and the second period, between M7 and M10 is OFF
  Interventions: Procedure: Deep brain Stimulation of cingulum anterior
- DBS-ACC OFF (Experimental): Start of stimulation of the DBS-ACC: On the first period, between M4 and M7, the DBS-ACC is OFF and the second period, between M7 and M10 is ON
  Interventions: Procedure: Deep brain Stimulation of cingulum anterior

INTERVENTIONS:
Procedure: Deep brain Stimulation of cingulum anterior — The Deep brain Stimulation of cingulum anterior is alternatively ON and OFF while Thalamic stimulation is ON

SUMMARY:
Deep brain stimulation (DBS) of the sensory thalamus has been proposed for 40 years to treat medically refractory neuropathic pain, but its efficacy remains partial and unpredictable. Recently, bilateral DBS of the dorsal anterior cingulate cortex (ACC), a brain region involved in the integration of the affective and cognitive aspects of pain, has been successively proposed to treat few patients suffering from refractory chronic pain, by decreasing the emotional impact of their chronic pain. ACC-DBS could be an alternative or complementary approach to thalamic DBS in these patients, but the consequences of chronic dACC-DBS on cognition and affects have not been studied specifically.

The primary objective is to evaluate the feasibility and safety of bilateral ACC-DBS combined with unilateral thalamic DBS in patients suffering from chronic unilateral pain, refractory to medical treatment. Secondary objective will evaluate the efficacy of this combined DBS compared to thalamic DBS only.

DETAILED DESCRIPTION:
Chronic pain represents a major personal and societal burden, especially for medically resistant patients. Deep brain stimulation (DBS) of the sensory thalamus has been proposed for 40 years to treat medically refractory neuropathic pain, but its efficacy remains partial and unpredictable. Recently, bilateral DBS of the dorsal anterior cingulate cortex (ACC), a brain region involved in the integration of the affective, emotional and cognitive aspects of pain, has been successively proposed to treat few patients suffering from refractory chronic pain. In a pilot study, 16 patients treated by ACC-DBS experienced a significant improvement of their quality of life despite a slight decrease of their pain intensity, by improving the affective and emotional impacts of their chronic pain. ACC-DBS could be an alternative or complementary approach to thalamic DBS in these patients. However the consequences of chronic dACC-DBS on cognition and affects have not been studied specifically.

The primary objective of this study is to evaluate the feasibility and safety of bilateral ACC-DBS combined with unilateral thalamic DBS in patients suffering from chronic unilateral pain, refractory to medical treatment. Secondary objective will evaluate the efficacy of this combined DBS compared to thalamic DBS only

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age 18-70 years old) suffering from chronic (duration >1 year) unilateral neuropathic pain
* severe (VAS score >6/10)
* with high emotional impact (HAD subscores > 10) considered as resistant to medication specific to neuropathic pain at sufficient doses and durations (including at least antiepileptics and antidepressants) and not sufficiently improved by rTMS and relevant surgical solutions.

Non inclusion criteria:

* previous history of stroke,
* cognitive impairment (MMSE score <24),
* DSMIV axis I psychiatric disorder,
* contra-indication to surgery, anesthesia or MRI;
* patient responder to rTMS,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-04-06 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Occurence of serious adverse events. | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  description of serious adverse events
Feasibility of ACC-DBS: success the process of surgical intervention | Day 0
  Feasibility of ACC-DBS will be evaluated by the proportion of patients undergoing with success the process of surgical intervention Safety will be evaluated by neurological examination
Feasibility of ACC-DBS : neurological success of the process of chronic stimulation | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  neurological success of the process of chronic stimulation will be evaluated by the neurological examination
Feasibility of ACC-DBS : psychiatric success of the process of chronic stimulation | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  psychiatric success of the process of chronic stimulation will be evaluated by the psychiatric assessment
Feasibility of ACC-DBS : cognitive success of the process of chronic stimulation | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  cognitive success of the process of chronic stimulation will be evaluated by the cognitive assessment

SECONDARY OUTCOMES:
Efficacy of ACC-DBS : change of pain intensity | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  Efficacy of ACC-DBS will be evaluated by pain intensity (VAS)
Efficacy of ACC-DBS : change of pain intensity | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  Efficacy of ACC-DBS will be evaluated by pain intensity (Brief Pain Inventory)
Efficacy of ACC-DBS : change of pain intensity | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  Efficacy of ACC-DBS will be evaluated by pain intensity (McGill Pain Questionnaire)
Efficacy of ACC-DBS : change of quality of life by SF-36 | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  Efficacy of ACC-DBS will be evaluated by quality of life (SF36).
Efficacy of ACC-DBS : change of quality of life by EQ-5D | Day 0, Month 1, Month 4, Month 7, Month 10, Month 22
  Efficacy of ACC-DBS will be evaluated by quality of life (EQ5D).

CONTACTS AND LOCATIONS:
Overall Officials: Denys FONTAINE, Principal Investigator — fontaine.d@chu-nice.fr
Locations (1):
- Department of neurosurgery, Nice, France

REFERENCES:
- [Derived] Fontaine D, Leplus A, Donnet A, Darmon N, Balossier A, Giordana B, Simonet B, Isan P, Regis J, Lanteri-Minet M. Safety and feasibility of deep brain stimulation of the anterior cingulate and thalamus in chronic refractory neuropathic pain: a pilot and randomized study. J Headache Pain. 2025 Feb 17;26(1):35. doi: 10.1186/s10194-025-01967-8. PMID 39962366
- [Derived] Leplus A, Isan P, Balossier A, Mouffok S, Donnet A, Papadopoulo T, Lanteri-Minet M, Regis J, Fontaine D. Somatotopy of the sensory thalamus: inputs from directional deep brain stimulation in pain patients. Ann Clin Transl Neurol. 2024 Jun;11(6):1502-1513. doi: 10.1002/acn3.52067. Epub 2024 Apr 26. PMID 38668642